CLINICAL TRIAL: NCT03185247
Title: Implementation of a Transdiagnostic Psychological Group Intervention for Pediatric Autonomic Dysfunction
Brief Title: Implementation of Transdx Group for POTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-0470
Record Dates: First submitted 2017-06-08; First posted 2017-06-14 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Dysautonomia; Anxiety; Depression
Keywords: Transdiagnostic; POTS (Postural Orthostatic Tachycardia Syndrome); Therapy
MeSH Terms: conditions — Autonomic Nervous System Diseases; Anxiety Disorders; Depression; Postural Orthostatic Tachycardia Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Intervention (Experimental): 10-week parent-child multi-family group
  Interventions: Behavioral: Transdiagnostic Group-Based Treatment

INTERVENTIONS:
Behavioral: Transdiagnostic Group-Based Treatment — 10 week 90-minute weekly therapy sessions including both the adolescent and caregiver. Treatment will consist of psychoeducation about dysautonomia, motivational interviewing techniques to promote readiness for change, support around lifestyle and behavioral changes, core CBT components (e.g., relaxation training, linking thoughts, feelings, and behaviors, minimizing catastrophizing thoughts, cognitive coping, and exposure), and components of ACT aiming to increase cognitive flexibility (e.g., mindfulness, experiential avoidance, values, cognitive defusion, committed action), and relapse prevention and maintenance. Most sessions will involve homework assigned to the adolescent and their parent/legal guardian(s) to encourage practice at home.

SUMMARY:
The proposed intervention is focused on developing and implementing a psychological approach incorporated into a group-based outpatient intervention for pediatric autonomic dysfunction. The investigators hypothesize that their intervention will result in improvements in the transdiagnostic mechanisms specifically targeted by components of their intervention including sleep, information processing, and youth/parent experiential avoidance.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent participants must be

  1. between the ages of 13-18 years old,
  2. english speaking, and
  3. have been diagnosed with autonomic dysfunction, dysautonomia, orthostatic intolerance, and/or POTS.
* Participants must also:

  1. endorse symptoms of autonomic dysfunction on the COMPASS 31 (measures are described below), and show
  2. moderate functional impairment, and/or
  3. some psychiatric symptoms in the domains of anxiety and/or depression.
* FDI scores must be greater than 12 (see Kashikar-Zuck et al., 2011 for an empirical rationale).
* Must have attended at least one day of school per week during the past month.
* On the measures of anxiety (SCARED) and depression (CDI), the adolescent's scale score must be above the "average" range based on T scores (CDI) or within the "clinical" range (SCARED).
* Each participant must have at least one English-speaking parent/legal guardian who can provide informed consent for the adolescent, as well as participate in the study.
* Each adolescent and their parent/legal guardian(s) must be English-speaking.

Exclusion Criteria:

* Adolescent participants;

  1. wards of the state,
  2. endorse active homicidal or suicidal ideation,
  3. have an intellectual disability, a pervasive developmental disability or significant developmental delay,
  4. endorse an active substance use disorder, and
  5. are currently participating in individual or group psychotherapy.
  6. do not have in-network health insurance that covers Health and Behavior interventions, or
  7. are unable to self-pay.
* Parent/legal guardian(s) are

  1. unwilling to participate in the study,
  2. are non-English speaking, or
  3. have an intellectual disability, a pervasive developmental disability or significant developmental delay, and/or
  4. do not have legal custody of the adolescent participant.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Composite Autonomic Symptom Score (self-report) | Baseline, 10 weeks, and 6-months
  This is a 31 item self-report measure developed to assess autonomic symptoms (e.g., dizziness, orthostatic intolerance, nausea, sweating).
Change in Functional Disability Inventory (caregiver and self-report) | Baseline, 10 weeks, and 6-months
  This is a measure that evaluates children's difficulty in physical and psychosocial functioning due to their physical health. The instrument consists of 15 items that assess self-perceptions of activity limitations during the past 2 weeks.
Change in Children's Depression Inventory (caregiver and self-report) | Baseline, 10 weeks, and 6-months
  This is a 27-item self-report measure designed to assess cognitive, behavioral, and affective symptoms of depression.
Change in Screen for Childhood Anxiety Related Emotional Disorders (caregiver and self-report) | Baseline, 10 weeks, and 6-months
  This measure is used to screen for childhood anxiety disorders including general anxiety disorder, separation anxiety disorder, panic disorder and social phobia. In addition, it assesses symptoms related to school refusal. The SCARED consists of 41 items.
Change in Transdiagnostic Youth/Parent Questionnaire | Baseline, 10 weeks, and 6-months
  Our team developed these comprehensive questionnaires to assess transdiagnostic mechanisms in the present study. These questionnaires comprise full measures and/or subscales drawn from several well-validated and psychometrically-sound measures that are available as part of the public domain and/or that were provided for open access by the developers of the measure, and that have been previously designed and validated to measure each of the mechanisms of interest. These mechanisms include emotion regulation, experiential avoidance, sleep, peer acceptance/rejection, parenting, and information processing.
Change in Pain Coping Questionnaire (caregiver and self-report) | Baseline, 10 weeks, and 6-months
  For the current study, this measure has been adapted to ask about "physical illness symptoms" rather than pain. The adapted measure asks adolescents/caregivers to indicate how often (1 = never to 5 = very often) they/their child used each of 39 coping strategies when responding to prompts such as, "When I am experiencing autonomic symptoms for a few hours or days, I…"
Satisfaction Questionnaire (caregiver and self-report) | 10 weeks
  This is an 8-item measure intended to assess satisfaction, perceived benefits, and likelihood of recommending the program. Items, which include "How would you rate the quality of care you have received?" are rated on a 1 to 4 Likert-scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Malmberg, PhD, Principal Investigator — University of Colorado/Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No